CLINICAL TRIAL: NCT02846649
Title: Feasibility and Acceptability of Using an Automated Text Messaging Program to Help Prevent Early Relapse Among Treatment-seeking Opioid Dependent Patients Discharged From the Emergency Department
Brief Title: A Text Messaging Program to Help Prevent Early Opioid Relapse
Acronym: PIER1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brian Suffoletto, MD, MS, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO15120183
Record Dates: First submitted 2016-07-06; First posted 2016-07-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PIER Intervention (Experimental): The program will help participants learn to recognize the presence of craving and how it can be reduced through environmental, self-regulatory and mood management. Each day, the PIER1 program sends (1) a morning reflection focused on positive thinking, (2) two random prompts assessing severity of craving, (3) feedback specific to managing withdrawal symptoms, mood management, and environmental triggers that are affecting craving, (4) evening assessments of drug use with feedback, (5) goal commitment prompt with feedback, and (6) user-triggered craving assessments with feedback
  Interventions: Behavioral: PIER

INTERVENTIONS:
Behavioral: PIER — Daily text message queries with tailored support

SUMMARY:
The objective is to determine feasibility and acceptability of a text message (SMS)-based relapse prevention intervention as measured through: (1) study retention and SMS query completion rates and (2) participant ratings of PIER1 interest, perceived efficacy, and ease of use. Methods: A mixed methods study of adult (age >=18) ED patients who seek treatment for opioids and have evidence of dependence based on Rapid Opioid Dependence Screen (RODS) score of >3 and are being discharged to outpatient (community) resources. All participants receive standard of care in the ED, complete a baseline web survey, are asked to text with us for at least 7 days (up to a max of 28 days) and are asked to complete a follow-up phone call between day 8 and 14. Investigators expect preliminary findings to support a relapse prevention intervention delivered through SMS. Based on feedback from this mixed methods study, investigators plan to test a refined SMS program in a randomized trial.

DETAILED DESCRIPTION:
The vast majority of those with opioid dependence do not receive treatment. This may be due to the limited availability of existing treatment programs and to a range of societal and individual-level barriers, including the stigma associated with identifying oneself as a substance user and difficulty attending a treatment program on a regular basis. Technology-based interventions have potential to help address these barriers and to expand access to evidence-based psychosocial treatment. Automated, computer-based interventions have found high user acceptance and utilization and shown promise in treating substance use disorders. The current study will evaluate a text-message-based psychosocial program called PIER1 (Preventing and Interrupting Early Relapse 1) when delivered to treatment-seeking opioid-dependent emergency department (ED) patients. PIER1 is an interactive program based on the Relapse Prevention Model. It is also informed by cognitive behavioral therapy and motivational interviewing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60 years
* Seeking treatment for substance abuse (chief complaint of "detox")
* English speaking
* Opioid dependence (nursing history of opioid use + RODS score>3)
* Ownership of a mobile phone with text messaging
* Medically and psychologically stable (as determined by the clinician or investigator)

Exclusion Criteria:

* No mobile phone ownership or mobile phone without text messaging capabilities
* Incarcerated/in police custody
* Being treated for a self-inflicted injury or suicidal ideation (as determined by the clinician)
* Medical condition affecting cognition (as determined by the clinician or investigator's discretion)
* Unable to read, speak, or comprehend English (at the clinician or investigator's discretion)
* Patients who are under the influence of illicit drugs or alcohol (at the clinician or investigator's discretion)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
SMS query completion rate | 7 days
  Investigators will report the percentage of SMS queries replied to over 7 days.

SECONDARY OUTCOMES:
Number of intentional opioid uses | 7 days
  Investigators will report the number of self-reported opioid use occasions.
Number of opioid overdoses | 7 days
  Investigators will report the number of self-reported opioid overdoses.
Ratings of usefulness | 7 days
  Investigators will report the median self-reported usefulness rating (0=not at all, 1=somewhat useful; 2=moderately useful; 3=very useful; 4=extremely useful

CONTACTS AND LOCATIONS:
Overall Officials: Brian Suffoletto, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Emergency Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will allow interested researchers access to a de-identified raw database